CLINICAL TRIAL: NCT00779779
Title: Reactogenicity and Safety of Two Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus Vaccine, Rotarix™ When Administered in Sri Lankan Infants Aged at Least 6 Weeks at the Time of First Vaccination.
Brief Title: Evaluation of Reactogenicity and Safety of GSK Biologicals' Rotarix™ (Human Rotavirus Vaccine) in Infants
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111664
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2010-07-30 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2011-02

CONDITIONS: Infections, Rotavirus
Keywords: Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — RIX4414 vaccine

GROUPS / COHORTS (1):
- Rotarix Group: Subjects received 2 oral doses of Rotarix vaccine at an interval of at least 4 weeks between doses. The first dose was given from the age of 6 weeks and vaccination with both doses was to be completed by 24 weeks of age.
  Interventions: Biological: Rotarix™

INTERVENTIONS:
Biological: Rotarix™ — Two oral doses, with at least 4 weeks interval in-between

SUMMARY:
This Post Marketing Surveillance (PMS) will collect reactogenicity and safety data on the use of human rotavirus vaccine in healthy infants aged from 6 weeks (first dose) to not more than 24 weeks (second dose).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol .
* A male or female at least 6 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.

Exclusion Criteria:

* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Any history of uncorrected congenital malformation of the gastrointestinal tract that would predispose for intussusception.
* Any contraindication as stated in the updated and approved Prescribing Information

Ages: 6 Weeks to 19 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 522 (Actual)
Dates: Start 2008-11-22; Primary Completion 2009-05-25 (Actual); Study Completion 2009-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Colombo, Sri Lanka

REFERENCES:
- [Background] Ruberu D et al. Post-marketing surveillance of a live-attenuated human rotavirus vaccine (Rotarix™) in India and Sri Lanka. Abstract presented at the 9th International Congress of Tropical Pediatrics (ICTP). Bangkok, Thailand, 18-20 October 2011.
- [Derived] Bravo L, Chitraka A, Liu A, Choudhury J, Kumar K, Berezo L, Cimafranca L, Chatterjee P, Garg P, Siriwardene P, Bernardo R, Mehta S, Balasubramanian S, Karkada N, Htay Han H. Reactogenicity and safety of the human rotavirus vaccine, Rotarix in The Philippines, Sri Lanka, and India: a post-marketing surveillance study. Hum Vaccin Immunother. 2014;10(8):2276-83. doi: 10.4161/hv.29280. PMID 25424932

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotarix Group
Started | 522
Completed | 498
Not Completed | 24
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 14
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Rotarix Group
Number analyzed (Participants) | 522
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 12.5 (5.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267
  Male | 255

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One >= Grade "2" Fever, Vomiting or Diarrhoea
Description: Grade 2 fever was defined as axillary temperature > 38.0 to <= 39.0 degrees Celsius and grade 3 fever as axillary temperature > 39.0 degrees Celsius.
  Grade 2 vomiting was defined as 2 episodes of vomiting per day and grade 3 as 3 or more episodes of vomiting per day.
  Grade 2 diarrhoea was defined as 4-5 looser than normal stools per day and grade 3 as 6 or more looser than normal stools a day.
Time Frame: During the 8-day solicited follow-up period
Population: Analysis was performed on the Total Vaccinated Cohort, which consisted of all vaccinated subjects with at least one vaccine administration documented.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 522
subjects | 78

2. Secondary Outcome: Number of Subjects Reporting Each Type of Solicited General Symptoms
Description: Solicited symptoms included cough, diarrhoea, irritability, loss of appetite, fever (degrees Celsius) and vomiting.
Time Frame: During the 8-day follow-up period
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 522
subjects
  Cough | 71
  Diarrhoea | 24
  Irritability | 124
  Loss of appetite | 83
  Fever | 152
  Vomiting | 45

3. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs cover any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day follow-up period
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 522
subjects | 25

4. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject
Time Frame: Throughout the study period (Day 0 to Month 3 or 4)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Rotarix Group
Number analyzed (Participants) | 522
subjects | 1

ADVERSE EVENTS:
Arm/Group | Rotarix Group
Serious Adverse Events (participants affected / at risk) | 1/522
Other Adverse Events (participants affected / at risk) | 247/522
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=522)
Crying (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4.6% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=522)
Cough (General disorders) | 71
Diarrhoea (General disorders) | 24
Loss of appetite (General disorders) | 83
Irritability (General disorders) | 124
Fever (General disorders) | 152
Vomiting (General disorders) | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.